CLINICAL TRIAL: NCT07137611
Title: Effect of Exercise Intensity on Neurochemical and Cognitive Function: The Role of Lactate and BDNF
Brief Title: Effects of Different Types of Exercise on BDNF and Cognitive Performance (Exercise-BDNF)
Acronym: Exercise-BDNF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, serkan pancar, Assoc. Prof., Aksaray University Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 01-121
Record Dates: First submitted 2025-06-25; First posted 2025-08-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Exercise Training; BDNF; Cognitive Functions; Lactate Blood Increase
Keywords: BDNF; exercise; cognitive function; trial making test; lactate
MeSH Terms: conditions — Hyperlactatemia; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low Intensity Exercise Group (n=3) (Experimental): They will be asked to perform low intensity exercise for the specified time, determined according to their maximal oxygen consumption capacity.
  Interventions: Behavioral: Low Exercise
- Moderate Intensity Exercise Group (n=3) (Experimental): They will be asked to perform moderate intensity exercise for the specified time, determined according to their maximal oxygen consumption capacity.
  Interventions: Behavioral: Moderate-Intensity Exercise
- High-Intensity Interval Training Group (n=3) (Experimental): They will be asked to perform HIIT exercise for the specified time, determined according to their maximal oxygen consumption capacity.
  Interventions: Behavioral: HIIT Exercise
- Control Group (n=3) (No Intervention): They will be asked to wait without exercising.

INTERVENTIONS:
Behavioral: Low Exercise — • Low-Intensity Continuous Training (LICT): Participants will run continuously for 24 minutes at 50-60% of their MAS without breaks.
  Other Names: Low Intensity Exercise
  Arms: Low Intensity Exercise Group (n=3)
Behavioral: Moderate-Intensity Exercise — Moderate-Intensity Continuous Training (MICT): Participants will run at a speed corresponding to 70-80% of their MAS. The protocol consists of four 4-minute bouts, separated by 2-minute active recovery periods, during which participants performed light jogging. This pattern totaled 24 minutes of exercise.
  Other Names: Moderate Intensity Exercise
  Arms: Moderate Intensity Exercise Group (n=3)
Behavioral: HIIT Exercise — High-Intensity Interval Training (HIIT): Participants will run at 110% of their MAS for 15-second intervals, covering a pre-calculated distance during each bout. After each 15-second sprint, they will rest passively for 15 seconds and returned to their starting point. This will be repeated continuously for 3 minutes, constituting one set. A total of four 3-minute sets will be completed, interspersed with 3-minute passive rest periods, yielding a total exercise time of 24 minutes.
  Arms: High-Intensity Interval Training Group (n=3)

SUMMARY:
Purpose The purpose of this study is to determine the acute effects of different exercise intensities (low, moderate, high) on brain-derived neurotrophic factor (BDNF) levels, trail making test performance, and perceived sensation scale.

Method

This randomized crossover controlled trial aimes to examine the acute effects of four experimental conditions-high-intensity interval training (HIIT), moderate-intensity continuous training (MICT), low-intensity continuous training (LICT), and a resting control (CTRL)-on cognitive performance (via the Stroop test, targeting executive function) and associated neurochemical responses (e.g., serum BDNF and blood lactate levels) in healthy young adults aged 18-25 years.

All participants will complete the four conditions in a randomized and counterbalanced manner. To ensure balanced exposure, they were assigned to one of four groups (n = 3 per group), each following a distinct condition order based on a Latin square design. This approach guaranteed that each session occurred equally across time points (sessions 1-4) and that the order minimized sequence effects by rotating the position of each condition relative to the others.

To control for potential carryover-particularly from elevated neurochemical responses following intense exercise (BDNF increases reported -no two high-intensity sessions will be scheduled consecutively. Where possible, higher and lower intensity protocols will be alternated. Furthermore, a seven-day interval separated each session to reduce residual physiological or cognitive effects.

The trial protocol was developed in line with CONSORT and SPIRIT guidelines, including relevant extensions for within-subject designs and non-pharmacological interventions. Participants were blinded to the study hypothesis (Pandis et al., 2017; Hopewell et al., 2025).

All exercise sessions will be conducted under supervision of a certified strength and conditioning coach to ensure consistency and adherence to protocol. in the morning (09:00-11:00) on a track and field pitch to control for chronobiological variation. Participants were instructed to avoid strenuous activity for 48 hours prior, abstain from alcohol and caffeine for 24 hours, and obtain at least 7-8 hours of sleep before each session. Dietary habits and general lifestyle were to remain unchanged throughout the study.

During the first visit, participants' body weight and body fat percentage were assessed using bioelectrical impedance analysis. Resting heart rate was then recorded, followed by administration of the Yo-Yo Intermittent Recovery Test Level 1 to determine maximal aerobic speed, aerobic capacity, and peak heart rate.

In the following four visits, each participant completed all experimental conditions. Each exercise session will begin with a standardized 10-minute warm-up, including light jogging, dynamic stretching, and movement preparation drills.

All exercise sessions were conducted on a standard track and field facility and lasted 40 minutes in total, consisting of a 10-minute standardized warm-up, 24 minutes of exercise, and a 5-minute recovery period. The exercise component was individually prescribed based on each participant's maximal aerobic speed, determined from the Yo-Yo Intermittent Recovery Test Level 1. All running distances were calculated individually using time × speed formulas based on each participant's maximal aerobic speed, ensuring workload equivalence across conditions.

* High-Intensity Interval Training: Participants ran at 110% of their MAS for 15-second intervals.
* Moderate-Intensity Continuous Training: Participants ran at a speed corresponding to 70-80% of their MAS.
* Low-Intensity Continuous Training: Participants ran continuously for 24 minutes at 50-60% of their MAS without breaks.
* Control: Participants remained seated at rest for the same duration (40 minutes), under the same environmental conditions and time schedule as the active conditions.

Venous blood samples were collected before and immediately after each session to assess neurochemical markers. Subsequently, cognitive performance was evaluated using the computerized Stroop test to measure executive function. Heart rate was continuously monitored during all exercise conditions using a Polar V800 device. Following each session, psychophysiological responses were assessed using the Rating of Perceived Exertion scale and the Exercise Enjoyment Scale.

ELIGIBILITY:
Inclusion Criteria

* Aged between 18 and 25 years
* No known medical condition that prevents participation in exercise
* Not currently using any pharmacological agents
* Exclusion Criteria:
* Experiencing any discomfort before, during, or after exercise
* Current or past diagnosis of pharmacological or doping substance use
* Engaging in regular exercise (more than 3 times per week) within the last 2 weeks
* History of alcohol or substance addiction
* Any other condition or factor that may prevent full participation in the study protocol

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male participants are eligible to participate in this study based on biological sex.
Enrollment: 12 (Actual)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
BDNF | Baseline and immediately after exercise (Day 1)
  BDNF will be measured using a Sunred brand ELISA kit from blood samples taken baseline and after exercise, and the results will be reported in pg/mL units.
Lactate | Baseline and immediately after exercise (Day 1)
  Lactate levels will be measured in millimoles per liter (mmol/L) from capillary/venous blood samples taken before and after exercise using a lactate analyzer.
Rating of Perceived Exertion Scale | Baseline and immediately after exercise (Day 1)
  Rating of Perceived Exertion (RPE) will be scored on the Borg 6-20 scale, where 6 indicates "no exertion" and 20 indicates "maximal exertion." Higher scores reflect greater perceived effort.
Exercise Enjoyment Scale | Baseline and immediately after exercise (Day 1)
  This outcome measures the participant's subjective enjoyment of the exercise session. Participants are asked to rate how much they enjoyed the exercise immediately after completion using a 7-point Likert scale ranging from 1 ("not enjoyable at all") to 7 ("extremely enjoyable"). The scale captures affective responses to physical activity, which can provide insight into adherence, motivation, and overall exercise experience.

CONTACTS AND LOCATIONS:
Overall Officials: serkan PANCAR, Assistant Professor, Study Director — Aksaray University /Faculty of Sports Sciences; Yakup Zühtü BİRİNCİ, Dr., Study Chair — Uludag Univesity
Locations (1):
- Aksaray University, Aksaray, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pandis N, Chung B, Scherer RW, Elbourne D, Altman DG. CONSORT 2010 statement: extension checklist for reporting within person randomised trials. Br J Dermatol. 2019 Mar;180(3):534-552. doi: 10.1111/bjd.17239. Epub 2019 Jan 4. PMID 30609010
- [Result] Hopewell S, Chan AW, Collins GS, Hrobjartsson A, Moher D, Schulz KF, Tunn R, Aggarwal R, Berkwits M, Berlin JA, Bhandari N, Butcher NJ, Campbell MK, Chidebe RCW, Elbourne D, Farmer A, Fergusson DA, Golub RM, Goodman SN, Hoffmann TC, Ioannidis JPA, Kahan BC, Knowles RL, Lamb SE, Lewis S, Loder E, Offringa M, Ravaud P, Richards DP, Rockhold FW, Schriger DL, Siegfried NL, Staniszewska S, Taylor RS, Thabane L, Torgerson D, Vohra S, White IR, Boutron I. CONSORT 2025 statement: updated guideline for reporting randomised trials. BMJ. 2025 Apr 14;389:e081123. doi: 10.1136/bmj-2024-081123. PMID 40228833
- See also: CONSORT 2025 statement: updated guideline for reporting randomised trials — https://pubmed.ncbi.nlm.nih.gov/40228833/
- See also: CONSORT 2010 statement: extension checklist for reporting within person randomised trials — https://pubmed.ncbi.nlm.nih.gov/30609010/